CLINICAL TRIAL: NCT05612334
Title: Randomized Controlled Study: Investigation of the Effect of Exercise on Liver Function Tests, Fatigue and Quality of Life in Patients With Liver Cirrhosis
Brief Title: Effect of Exercise on Liver Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HULYA KESKIN (Other)
Responsible Party: Sponsor-Investigator, HULYA KESKIN, Asst. Prof., Mardin Artuklu University
Organization: Mardin Artuklu University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EGE UNIVERSTIY
Record Dates: First submitted 2022-10-27; First posted 2022-11-10 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Liver Function Tests
Keywords: Liver Function Tests; Liver Cirrhosis; Exercise; Fatigue; Quality of Life
MeSH Terms: conditions — Liver Cirrhosis; Motor Activity; Fatigue | interventions — Exercise; Breathing Exercises

STUDY DESIGN:
Intervention Model Description: First, they were informed about the benefits of exercise and walking. They were also informed about the duration and type of exercise and what should be considered before, during, and after exercises. Then, an informative training booklet prepared by the researcher containing the same information was given to them. An exercise program (5 minutes warm-up-30 minutes walking-5 minutes cooling down) was demonstrated to the patient by the researcher, and then the patient performed the first exercise under the supervision of the researcher. Beginning with the second exercise, the patient performed a 40-minute exercise program, 3 days a week, for 3 months. During this period, the researcher regularly made phone calls once a week to motivate the patient and check whether the patient performed the exercise program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental (Experimental): The data collection forms used in the research were applied in the treatment group at the first polyclinic visit (0. month) via face-to-face interviews. First, they were informed about the benefits of exercise and walking. They were also informed about the duration and type of exercise and what should be considered before, during, and after exercises. Then, an informative training booklet prepared by the researcher containing the same information was given to them. An exercise program (5 minutes warm-up-30 minutes walking-5 minutes cooling down) was demonstrated to the patient by the researcher, and then the patient performed the first exercise under the supervision of the researcher. Beginning with the second exercise, the patient performed a 40-minute exercise program, 3 days a week, for 3 months. During this period, the researcher regularly made phone calls once a week to motivate the patient and check whether the patient performed the exercise program.
  Interventions: Behavioral: exercise (5 minutes warm-up-30 minutes walking-5 minutes cooling down)
- Placebo (Placebo Comparator): The breathing exercise group, which constitutes the placebo-control group, was first informed about correct breathing techniques by the researcher, and an informative training brochure prepared by the researcher, containing correct breathing exercise information, was given to them. The exercise was performed by the researcher and shown to the patient. The first exercise was performed by the patient under the supervision of the researcher. They were informed about the continuation of the breathing exercise program for 3 months, once a day for 10 minutes, starting from the 2nd exercise. Regular phone calls were made once a week.
  Interventions: Behavioral: exercise (5 minutes warm-up-30 minutes walking-5 minutes cooling down)
- No intervention (No Intervention): The control group was contacted by regular phone calls once a week to monitor their compliance with the treatment, to encourage them to express their problems, if any, and to motivate them for the treatment process.

INTERVENTIONS:
Behavioral: exercise (5 minutes warm-up-30 minutes walking-5 minutes cooling down) — the breathing exercise group, which constituted the placebo control group, were first informed by the researcher about the correct breathing techniques and was given an informative training brochure prepared by the researcher containing the correct breathing exercise information.
  Other Names: Behavioral; breathing exercise
  Arms: Experimental; Placebo

SUMMARY:
This randomized controlled study aimed to determine the effect of the exercise program to be applied in patients with cirrhosis on the patient's biochemistry parameters, quality of life, fatigue level, depression, and sleep quality.

DETAILED DESCRIPTION:
This randomized controlled study aimed to determine the effect of the exercise program to be applied in patients with liver cirrhosis on the patient's biochemistry parameters, quality of life, fatigue level, depression, and sleep quality. The universe of the study consisted of patients with stage I and II liver cirrhosis according to Child-Pugh A and B scores followed-up in Ege University Faculty of Medicine Hospital Gastroenterology Department Hepatology Polyclinic. The sample of the study consisted of a total of 90 patients, including 30 patients in the intervention group, 30 patients in the control group, and 30 patients in the placebo-control group (n=90). The study was completed with a total of 84 patients, including the intervention group (n=27), the control group (n=28), and the placebo control group (n=29). The data collection stage of the study was carried out between August 20, 2019 and March 04, 2020. The data collection forms used in the study were applied to the exercise intervention group at the first polyclinic visit (0th month) by face-to-face interview method. An exercise program (5 minutes warm-up, 30 minutes walking, 5 minutes cooldown) was demonstrated to the patient by the researcher, a booklet containing the exercise information prepared by the researcher was given, and the patient performed the first exercise under the supervision of the researcher. The patient followed a 40-minute exercise program, 3 days a week, for 3 months on his/her own starting from the second exercise. The researcher regularly made motivating and encouraging phone calls to the patient with phone follow-up once a week and also checked whether the patient followed the exercise program during this period. Similarly, the breathing exercise group, which constituted the placebo control group, were first informed by the researcher about the correct breathing techniques and was given an informative training brochure prepared by the researcher containing the correct breathing exercise information. Regularly, the control group was contacted only once a week to check the patients' compliance with the treatment, to encourage them to express their problems, if any, and to motivate them for the treatment process. The forms used to collect the research data were Personal Information Form, 6-Minute Walking Test, Body Mass Index Assessment Form, SF-36 Quality of Life Scale, Biochemistry Parameters Assessment Form, Child-Pugh Score Assessment Form, Beck's Depression Inventory, Fatigue Severity Scale, Pittsburgh Sleep Quality Index (PSQI), and these were applied to the patients by face-to-face interview method. Data collection forms other than Personal Information Form were applied twice at the beginning of the study and the end of the 12th week. Statistical analyses were performed using IBM SPSS Statistics 25.0 (IBM SPSS Statistics for Windows, Version 25.0. Armonk, NY: IBM Corp.). Descriptive statistics of the data were given as mean, standard deviation, median, minimum, maximum, frequency, and percentage values. The assumption of normality of quantitative data was checked by the Shapiro-Wilk test. For the case in which the assumption of normality was not met, the non-parametric Brunner-Langer model was tested using the R 4.0.2 software (R software, version 4.0.2, package: nparLD, R Foundation for Statistical Computing, Vienna, Austria; http://r-project.org) in numerical data using the 'group effect', 'time effect', and 'group-time interaction' (F1-LD-F1 design).

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years old and over
* Cirrhosis of Stage I or Stage II results (Child pugh A: 5-6 (good) compensated disease) -B:7-9 Serious clinical clinical)
* Absence of specific musculoskeletal limitations (history of arthritis, joint swelling)
* No history of falls (≥3 falls in the past year)
* Absence of advanced cerebrovascular and peripheral vascular insufficiency
* Willingness to participate in the study

Exclusion Criteria:

* Be younger than 18 years old
* Child pugh C diagnosed with stage III or stage IV liver cirrhosis
* Platelet <20.000mm3/blood
* Hemoglobin <8 g/dl
* Heart rate <50 or >100
* Blood pressure systolic >160 mmHg and diastolic >85 mmHg
* 0xygen saturation <92%
* Specific musculoskeletal limitations (history of arthritis, joint swelling)
* History of falls (≥3 falls in the past year)
* Blood glucose below 70 mg/dl
* Uncontrollable metabolic disease
* Presence of advanced cerebrovascular and peripheral vascular insufficiency
* Not being willing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Information Form | 10 minutes
  The Information Form, developed by the researcher in line with the literature, consists of 15 items inquiring about age, gender, marital status, education status, health insurance, occupation, smoking and alcohol use, drugs used, presence of concomitant diseases, cirrhosis etiology, duration since diagnosis, and disease stage.
6-Minute Walk Test (6-MWT) | 6 minutes
  It is a test used in the follow-up of chronic cardio-pulmonary diseases and in the reliable evaluation of functional performance. It is based on the patient's walking for 6 minutes along a corridor, usually 30 meters long, with marked start and end points
Body Mass Index Evaluation Form | 3 minutes
  It is a form in which weight, height, and thigh circumference measurements of the patients were recorded at follow-up months 0, 2, and 3.
SF-36 Quality of Life Scale | 10 minutes
  It is among the general scales commonly used to measure quality of life.
Biochemistry Parameters Evaluation Form | 5 minutes
  It is the form that includes information, collected at the 1st and 12th weeks, about the follow-up of laboratory tests such as AST, ALT, GGT, ALP, LDH, Total Protein, Albumin, Total Bilirubin, and Direct Bilirubin, which is called the liver function tests performed in the routine outpatient clinic controls of patients with liver cirrhosis.
Child-Pugh Score Evaluation Form | 7 minutes
  Child class is associated with the likelihood of developing complications of cirrhosis. For example, patients with Child class C cirrhosis are more likely to have variceal bleeding than those with class A cirrhosis.
Beck Depression Inventory | 10 minutes
  It was developed by Beck et al. in 1961 to measure the behavioral manifestations of depression in adolescents and adults, and its validity and reliability study in Turkey was performed by Hisli (Beck et al., 2015)(Hisli, 1989). Patients were asked to mark their status for the last week, including the then-current day. It consists of 21 items related to depressive symptoms such as guilt, pessimism, sense of failure, dissatisfaction, fatigue, sleep, and appetite, and each item is scored between 0 and 3. An increased score indicates that the severity of depression is higher. The total score is 63. According to this scale, 1-10 points are considered normal, 11-16 points indicate mild mental distress, 17-20 points indicate borderline clinical depression, 21-30 points indicate moderate depression, 31-40 points indicate severe depression, and above 40 points indicate very severe depression (Hisli, 1989).
Fatigue Severity Scale | 10 minutes
  The Fatigue Severity Scale, which is used to evaluate the level of fatigue, was developed by Krupp et al., and its Turkish validity and reliability were verified by Armutlu et al. (Annex XIII). The scale consists of 9 items, and each item is scored as 1 (strongly disagree) - 7 (totally agree). The total score of the scale is the average of the value given to all questions. A high score indicates increased fatigue severity. An average score of 4 or above indicates severe fatigue (Krupp et al., 1989)(Armutlu et al., 2007).
Pittsburgh Sleep Quality Index (PSQI) | 10 minutes
  The Pittsburg Sleep Quality Index (PSQI) is a 19-item self-report scale that evaluates sleep quality and disorder, and was developed by Buysse et al. in 1989. Turkish validity and reliability was established by Ağargün et al. (Buysse et al., 1989)(Ağargün, 1996). The questionnaire consists of 18 items and 7 components (subjective sleep quality, sleep duration, sleep disturbance, sleep latency, habitual sleep efficiency, sleep medication use, and daytime dysfunction). Score of each component is calculated by taking into account the scores obtained from the related items. In line with these questions, information about the frequency, severity, and sleep latency of the person's sleep-related problems is obtained. The total score is obtained by summing up the 7 components. A total score of 0-21 is obtained. A score greater than 5 indicates poor sleep quality. An increase in the score indicates deterioration in sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: HÜLYA KESKİN, Principal Investigator — Mardin Artuklu University, Faculty of Health Science
Locations (1):
- Hülya Keskin, Mardin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The study can be reviewed by other researchers after the study has been published.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: data will be shared as long as they are published
Access Criteria: publication page